CLINICAL TRIAL: NCT00595374
Title: Efficacy and Safety Comparison of Insulin Detemir Plus Insulin Aspart to Insulin NPH Plus Insulin Aspart in Adults With Type 1 Diabetes Mellitus
Brief Title: Efficacy and Safety of Insulin Detemir in Type 1 Diabetes
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NN304-1582
Record Dates: First submitted 2008-01-07; First posted 2008-01-16 (Estimated); Last update posted 2017-02-24 (Actual); Status verified 2017-02

CONDITIONS: Diabetes; Diabetes Mellitus, Type 1
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 1 | interventions — Insulin Detemir; Insulin, Isophane; Insulin Aspart

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: insulin detemir
Drug: insulin NPH
Drug: insulin aspart

SUMMARY:
This trial is conducted in Europe.

The aim of this trial is to compare the efficacy and safety of insulin detemir and insulin NPH in adults with type 1 diabetes on blood glucose control.

ELIGIBILITY:
Inclusion Criteria:

* Duration of type 1 diabetes for at least 12 months
* BMI below 35 kg/m2
* HbA1c between 7.0-12.0%
* Current treatment with preprandial short acting insulin and insulin NPH once or twice daily for at least 6 months
* Fertile females must use acceptable method of contraception if there is any risk of pregnancy in the opinion of the Investigator

Exclusion Criteria:

* Known or suspected allergy to trial product or related products
* Previous participation in this trial
* Receipt of any investigational products within the last 2 months prior to this trial
* Drug or alcohol dependence
* Pregnancy, breast-feeding or intention of becoming pregnant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 114 (Actual)
Dates: Start 2003-12-02 (Actual); Primary Completion 2004-10-07 (Actual); Study Completion 2004-10-07 (Actual)

PRIMARY OUTCOMES:
HbA1c | after 26 weeks of treatment

SECONDARY OUTCOMES:
Plasma glucose profiles
Change in body weight
Quality of Life
Incidence of adverse events
Incidence of hypoglycaemic episodes

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (17):
- Netherlands (17):
  - Novo Nordisk Investigational Site, Amersfoort
  - Novo Nordisk Investigational Site, Apeldoorn
  - Novo Nordisk Investigational Site, Den Helder
  - Novo Nordisk Investigational Site, Deventer
  - Novo Nordisk Investigational Site, Enschede
  - Novo Nordisk Investigational Site, Gouda
  - Novo Nordisk Investigational Site, Hoogeveen
  - Novo Nordisk Investigational Site, Leidschendam
  - Novo Nordisk Investigational Site, Meppel
  - Novo Nordisk Investigational Site, Rotterdam
  - Novo Nordisk Investigational Site, Stadskanaal
  - Novo Nordisk Investigational Site, The Hague
  - Novo Nordisk Investigational Site, Utrecht
  - Novo Nordisk Investigational Site, Waalwijk
  - Novo Nordisk Investigational Site, Weert
  - Novo Nordisk Investigational Site, Zevenaar
  - Novo Nordisk Investigational Site, Zwolle

REFERENCES:
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com